CLINICAL TRIAL: NCT06327178
Title: Response to the Combination of Stereotactic Body Radiation Therapy and Concurrent PD-1 Blockade in Patients With Metastatic Renal Cell Carcinoma: a Retrospective Study
Brief Title: Systemic Anti-tumor Activity and Safety of the Combination of SBRT and Concurrent PD-1 Blockade in Metastatic RCC.
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-520
Record Dates: First submitted 2024-03-11; First posted 2024-03-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Systemic Anti-tumor Activity and Safety of the Combination of SBRT and Concurrent PD-1 Blockade in Metastatic RCC
Keywords: stereotactic body radiotherapy, abscopal effects; PD-1 blockade

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prior research has indicated that stereotactic body radiotherapy (SBRT) can effectively trigger systemic anti-tumor immune response. The goal of this observational study is to learn about abscopal effects of stereotactic body radiotherapy and concurrent anti-PD-1 antibody treatment in patients of metastatic clear renal cell carcinoma. The primary objective was to assess the objective response rate (ORR) in non-irradiated lesions, and incidence of adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years at the time of signing informed consent;
* Histologically confirmed, advanced renal cell carcinoma of stage IV (AJCC 8);
* Previously received SBRT and concurrent PD-1 blockade treatment；
* Evidence of measurable metastatic kidney cancer according to RECIST 1.1 criteria.

Exclusion Criteria:

* Patients who cannot be adequately followed up;
* Has a known additional malignancy that is progressing or requires active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced metastatic clear cell renal cell carcinoma who have received SBRT and concurrent PD-1 blockade treatment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China